CLINICAL TRIAL: NCT02759341
Title: Tako-Tsubo Cardiomyopathy and Cardiac Syndrome X: a Study on the Brain-heart Interactions in Two Orphan Cardiac Diseases.
Brief Title: Brain-heart Interactions in Tako-Tsubo Cardiomyopathy and Cardiac Syndrome X:
Acronym: BRAINHEART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale San Giovanni Bellinzona (Other)
Collaborators: Swiss Heart Foundation (Other)
Responsible Party: Principal Investigator, Mattia Cattaneo, M.D., Ospedale San Giovanni Bellinzona
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CE 3015; 2016-00015 (Other: Swissethic)
Record Dates: First submitted 2016-04-25; First posted 2016-05-03 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Takotsubo Cardiomyopathy; Cardiac X Syndrome; Acute Myocardial Infarction
MeSH Terms: conditions — Takotsubo Cardiomyopathy; Microvascular Angina

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cardiac X Syndrome (CSX) (Other): patients with Cardiac X Syndrome (CSX), according to the diagnostic criteria previously proposed by Lanza (Lanza, Heart. 2007)
  Interventions: Other: Manual for the Assessment and Documentation of Psychopathology (AMDP 8); Other: Million Clinical Multiaxial Inventory 3 (MCMI-III); Other: State-Trait Anxiety Inventory form Y (STAI-Y); Other: SF-36 Health-Related Quality of Life; Other: Blood oxygenation level dependent- functional Magnetic Resonance Imaging (BOLD-fMRI)
- Takotsubo Cardiomyopathy (TTC) (Other): Tako-Tsubo Cardiomyopathy (TTC), according to Mayo diagnostic criteria at least six months after the event. (Prasad A, et al. Am Heart J. 2008)
  Interventions: Other: Manual for the Assessment and Documentation of Psychopathology (AMDP 8); Other: Million Clinical Multiaxial Inventory 3 (MCMI-III); Other: State-Trait Anxiety Inventory form Y (STAI-Y); Other: SF-36 Health-Related Quality of Life; Other: Blood oxygenation level dependent- functional Magnetic Resonance Imaging (BOLD-fMRI)
- Acute myocardial infarction (AMI) (Other): Type 1, 4a, 4b myocardial infarction (ST-segment elevation acute myocardial infarction [STEMI] and Non ST-segment elevation acute myocardial infarction [NSTEMI] acute coronary syndrome [ACS] with significant ≥70% coronary stenosis) at least six months after the event. (Thygesen K, et al. Eur Heart J. 2012)
  Interventions: Other: Manual for the Assessment and Documentation of Psychopathology (AMDP 8); Other: Million Clinical Multiaxial Inventory 3 (MCMI-III); Other: State-Trait Anxiety Inventory form Y (STAI-Y); Other: SF-36 Health-Related Quality of Life; Other: Blood oxygenation level dependent- functional Magnetic Resonance Imaging (BOLD-fMRI)

INTERVENTIONS:
Other: Manual for the Assessment and Documentation of Psychopathology (AMDP 8)
Other: Million Clinical Multiaxial Inventory 3 (MCMI-III)
Other: State-Trait Anxiety Inventory form Y (STAI-Y)
Other: SF-36 Health-Related Quality of Life
Other: Blood oxygenation level dependent- functional Magnetic Resonance Imaging (BOLD-fMRI)

SUMMARY:
The Tako-Tsubo Cardiomyopathy (TTC) and the Cardiac Syndrome X (CSX) are respectively acute and chronic heart diseases, which mimic myocardial infarction and stable angina pectoris without alterations of large coronary vessels. The causes and the most appropriate and best treatment for these diseases have not been yet clarified, but there are indications, that mental and psychosocial aspects may also contribute to these two diseases. So far, there is no study, which has comprehensively evaluated the interactions between mind and heart in these two conditions.

The purpose of this study is to search for possible differences in mental activity, response to stressful events and function of specific areas of the brain deeply involved in relation between mind and heart.

45 subjects will be recruited and divided equally into: patients with CSX, patients with TTC (at least 6 months ago) and patients with previous acute myocardial infarction (at least 6 months ago). All participants will undergo a clinical interview and several questionnaires that assess various mental functions, the stress response and the quality of life. In addition, in a separate visit the participants will undergo a Magnetic Resonance Imaging without contrast medium that helps to assess function of specific areas of the brain.

ELIGIBILITY:
Inclusion Criteria:

* Group A. 15 patients with Cardiac X Syndrome (CSX), according to the diagnostic criteria previously proposed by Lanza et al.
* Group B. 15 patients with Tako-Tsubo Cardiomyopathy (TTC), according to Mayo diagnostic criteria at least 6 months after being hospitalized or diagnosed with TTC.
* Group C (control group). 15 prospectively enrolled patients with previous Type 1, 4a, 4b myocardial infarction (ST-segment elevation acute myocardial infarction [STEMI] and Non ST-segment elevation acute myocardial infarction [NSTEMI] acute coronary syndrome [ACS] with significant ≥70% coronary stenosis) at least six months after the event.

Acute myocardial infarction will be defined according to the third universal definition of myocardial infarction.

Exclusion Criteria:

* Refused consent
* Unable to participate or provide written informed consent
* Short-term survival (<1 year)
* Acute or decompensated medical conditions
* Acute neurological or psychiatric diseases
* Absence of sinus rhythm or frequent ectopic beats
* History of severe lung, liver, kidney or autoimmune diseases
* Any contraindication to MRI

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-02; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Difference in BOLD-fMRI intensity signal in CSX and TTC as compared to AMI patients | Baseline
Difference in BOLD-fMRI distribution signal in CSX and TTC as compared to AMI patients | Baseline

SECONDARY OUTCOMES:
Difference in CSX and TTC AMDP 8 results as compared to AMI patients | Baseline
Difference in CSX and TTC MCMI-III results as compared to AMI patients | Baseline
Difference in CSX and TTC STAI-Y results as compared to AMI patients | Baseline
Difference in CSX and TTC SF-36 HRQOL results as compared to AMI patients | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mattia Cattaneo, MD, Principal Investigator — Ospedale San Giovanni Bellinzona; Augusto Gallino, MD, Study Chair — Ospedale San Giovanni Bellinzona
Locations (1):
- Ospedale Regionale di Bellinzona e Valli - Ospedale San Giovanni Bellinzona, Bellinzona, Canton Ticino, Switzerland

REFERENCES:
- [Background] Lanza GA. Cardiac syndrome X: a critical overview and future perspectives. Heart. 2007 Feb;93(2):159-66. doi: 10.1136/hrt.2005.067330. Epub 2006 Jan 6. PMID 16399854
- [Background] Prasad A, Lerman A, Rihal CS. Apical ballooning syndrome (Tako-Tsubo or stress cardiomyopathy): a mimic of acute myocardial infarction. Am Heart J. 2008 Mar;155(3):408-17. doi: 10.1016/j.ahj.2007.11.008. Epub 2008 Jan 31. PMID 18294473
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Writing Group on the Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Thygesen K, Alpert JS, White HD, Jaffe AS, Katus HA, Apple FS, Lindahl B, Morrow DA, Chaitman BA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S; ESC Committee for Practice Guidelines (CPG). Third universal definition of myocardial infarction. Eur Heart J. 2012 Oct;33(20):2551-67. doi: 10.1093/eurheartj/ehs184. Epub 2012 Aug 24. No abstract available. PMID 22922414
- [Derived] Cattaneo MM, Pravata E, Provenzi M, Moccetti M, Kaelin A, Sudano I, Biasucci L, Gallino C, Limoni C, Calanchini C, Gallino A, Crea F, Cattaneo M. Role of the central autonomic nervous system intrinsic functional organisation and psychosocial factors in primary microvascular angina and Takotsubo syndrome. Open Heart. 2020 Jul;7(2):e001315. doi: 10.1136/openhrt-2020-001315. PMID 32727853